## SAFE at Home: A Service to Provide Social Engagement to Community-Dwelling Persons With Dementia NCT05516147

Statistical Analysis Plan 12/1/23

The SAFE at Home app will be considered successful if persons with dementia exhibit higher levels of positive engagement/affect and lower levels of negative engagement- as measured by the Menorah Park Engagement Scale (MPES)-during the intervention, as compared to known means for standard programming. Multiple observations of participants will be taken during SAFE at Home programming. Then, means will be calculated for each participant for each item (on the MPES) or positive and negative subscale (for the EPWDS). Then, we will conduct a one-sample *t*-test to determine whether there are significant differences between the known means and the means observed during SAFE at Home programming. We will also conduct paired sample *t*-tests to examine whether participants exhibit an improvement in the Dementia-Related Quality of Life Scale (DEMQOL), Geriatric Depression Scale – Short Form (GDS-SF), Neuropsychiatric Inventory – Nursing Home (NPI-NH), and the UCLA Loneliness Scale (ULS).